CLINICAL TRIAL: NCT03510507
Title: Characteristics of Positive Lyme PCR Arthritis, Data From CNR Borrelia 2011-2016
Brief Title: Characteristics of Lyme Arthritis
Acronym: ArthLyme
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6971
Record Dates: First submitted 2018-02-26; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-01

CONDITIONS: Lyme Arthritis
Keywords: Lyme arthritis; Borrelia burgdorferi; vector tick; Arthritis; joints
MeSH Terms: conditions — Lyme Disease; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lyme disease is due to Borrelia burgdorferi sensu lato and is transmitted by a tick vector of the genus Ixodes. One of the clinical forms of this disease in the disseminated phase is the appearance of arthritis, classically mono or oligo-arthritis in the large joints.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of Lyme arthritis confirmed by PCR of joint fluid at CNR Borrelia between 2011 and 2016
* Patient who has agreed to use his medical data for research purposes

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with Lyme arthritis and confirmed by PCR of joint fluid at CNR Borrelia between 2011 and 2016
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of clinical and biological data of French patients with Lyme arthritis between 2011 and 2016 | The period from 2011 to 2016 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Benoit JAULHAC, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Laboratoire de Bacteriologie - Ptm, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No